CLINICAL TRIAL: NCT04811651
Title: Umbilical Cord-derived Mesenchymal Stem Cells for Ischemic Stroke (UMSIS): a Prospective, Double-blinded, Randomized Controlled, Pilot Study
Brief Title: Umbilical Cord-derived Mesenchymal Stem Cells for Ischemic Stroke
Acronym: UMSIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Director of neurology department, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: k（2019）46
Record Dates: First submitted 2021-03-15; First posted 2021-03-23 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Ischemic Stroke
Keywords: Ischemic Stroke; Stem Cell
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Two different treatment groups; intravenous umbilical cord-derived mesenchymal stem cells or intravenous placebo solution
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Treatment and placebo solutions have identical appearance. Protocols will be designed to ensure that the physician evaluating patient safety and efficacy outcome as well as laboratory analysis, will not have access to the randomisation codes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): intravenous umbilical cord derived mesenchymal stem cells
  Interventions: Biological: Umbilical Cord-derived Mesenchymal Stem Cells
- Placebo Comparator (Placebo Comparator): intravenous placebo solution with the same appearance as the treatment group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Umbilical Cord-derived Mesenchymal Stem Cells — umbilical cord derived mesenchymal stem cells were intravenously injected in a single dose of one hundred million.
  Arms: Treatment group
Drug: Placebo — intravenous placebo solution with the same appearance as the treatment group.
  Arms: Placebo Comparator

SUMMARY:
This is a doble blind, placebo controlled clinical trial to assess safety and efficacy of intravenous administration of Umbilical cord-derived Mesenchymal Stem cells in patients with ischemic stroke within 6 months of onset.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-80 years old;
2. Patients with anterior circulation cerebral infarction;
3. NIHSS: 6-25, and the limb movement score is at least 2 points;
4. Hemoglobin > 115g / L, platelet > 100 × 109 / L, leukocyte > 3 × 109 / L;
5. the time from onset to treatment: group A（6-24 hours）、group B（1-3 days）、gourp C（4-7 days）、group D（1-4 weeks）、group E（1-6 months）;
6. The patient or the legal representative of the patient can and is willing to sign the informed consent.

Exclusion Criteria:

1. Patients who need or expect decompressive craniectomy;
2. Patients who need or are expected to receive endovascular treatment ;
3. Patients receiving intravenous thrombolysis;
4. Disturbance of consciousness；
5. Pregnant women or women of childbearing age who have not taken effective contraceptive measures;
6. Intracranial hemorrhagic diseases: cerebral hemorrhage, subarachnoid hemorrhage, etc;
7. Posterior circulation cerebral infarction;
8. Tumor patients;
9. Epilepsy patients;
10. Severe neurological deficit caused by stroke (MRS = 5);
11. Previous diseases with obvious functional impairment, such as Parkinson's disease, motor neuron disease, moderate Alzheimer's disease, osteoarthritis, etc;
12. Patients with history of coagulation disorders, systemic bleeding tendency and thrombocytopenia (< 100000 / mm3);
13. Chronic liver disease, liver and kidney dysfunction, elevated ALT or ast (2 times higher than the upper limit of normal value), elevated serum creatinine (1.5 times higher than the upper limit of normal value) or dependent on renal dialysis;
14. Patients with moderate to severe mental illness obviously interfere with treatment compliance;
15. Patients with high blood pressure (systolic blood pressure > 180mmhg) or low blood pressure (systolic blood pressure < 90mmHg);
16. The expected survival time is less than one year;
17. Those who have conducted other trials within 3 months;
18. Other circumstances considered unsuitable by the researcher.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Proportion of modified Rankin Scale (mRS) 0-2 | 90 Days
  the minimum and maximum values of mRS are 0 and 6, respectively; higher mRS mean a worse outcome

SECONDARY OUTCOMES:
Proportion of modified Rankin Scale (mRS) 0-2 | 180，360 Days
  the minimum and maximum values of mRS are 0 and 6, respectively; higher mRS mean a worse outcome
changes in Fugl-Meyer scale | 90days；180days；360days
  Fugl-Meyer Assessment Scale ranges from 0 to 100.
changes in Purdue hand function test | 90days；180days；360days
  The changes of fine motor function were evaluated by Purdue hand function test
changes in box and block test | 90days；180days；360days
  The changes of fine motor function were evaluated by box and block test
Proportion of modified Rankin Scale (mRS) 0-1 | 90days；180days；360days
  the minimum and maximum values of mRS are 0 and 6, respectively; higher mRS
changes in the national institutes of health stroke scale (NIHSS) | 90days；180days；360days
  NIHSS ranges from 0-42, and high NIHSS means bad outcome
changes in Mini-mental State Examination (MMSE) score | 90days；180days；360days
  MMSE score ranges from 0 to 30.
changes in Montreal Cognitive Assessment (MoCA) score | 90days；180days；360days
  MOCA score ranges from 0 to 30.
The changes of head images | 90days；180days；360days
  head images included flair, DTI
changes in some serum biomarkers | 90days；180days；360days
  serum biomarkers included CPEC, VEGF, BDNF, MMP-9

OTHER OUTCOMES:
Number of Adverse Events | 360days

CONTACTS AND LOCATIONS:
Overall Officials: Chen Hui-Sheng, Doctor, Principal Investigator — General Hospital of Shenyang Military Region
Locations (1):
- Department of Neurology, General Hospital of Northern Theater Command, Shenyang, China